CLINICAL TRIAL: NCT02568904
Title: The Effects of Binge Drinking on Innate Host Defence Mechanisms
Brief Title: Alcohol and Innate Immunity
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Alcohol01
Record Dates: First submitted 2015-07-29; First posted 2015-10-06 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Binge Drinking
MeSH Terms: conditions — Binge Drinking | interventions — Ethanol; Glucose; Fructose

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Urine, Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Alcohol binge: Healthy volunteers receive 2ml vodka 40% per kg bodyweight as a binge
  Interventions: Other: Alcohol
- Fructose: 75 g Fructose orally
  Interventions: Other: Fructose
- Glucose: 75 g Glucose orally
  Interventions: Other: Glucose
- Vehicle: 2ml tap water per kg body weight
  Interventions: Other: vehicle

INTERVENTIONS:
Other: Alcohol — every participant will drink vodka at a dose of 2ml/kg bodyweight
  Groups: Alcohol binge
Other: Glucose — oral Glucose tolerance test
  Groups: Glucose
Other: Fructose — oral fructose tolerance test
  Groups: Fructose
Other: vehicle — control (water)
  Groups: Vehicle

SUMMARY:
Alcohol leads to a leaky gut and translocation of bacterial products. This may lead to inflammation and immune dysfunction as well as the typical hangover symptoms.

DETAILED DESCRIPTION:
Alcohol binge drinking, defined as 5 or more drinks for men and 4 or more drinks for women at one time, is the most frequent form of alcohol consumption worldwide, especially in younger people. This drinking pattern is popular and leads to increased mortality and morbidity. Therefore binge drinking is a major public health issue. The behavioural and neurological consequences of binge drinking are well characterized.

Less is known about the systemic effects on the gut as the first organ in contact with alcohol. Chronic alcohol intake can lead to increased gut permeability, bacterial translocation and alterations in the gut microbiome in animal models. Recently bacterial translocation has been shown in healthy volunteers after a single alcohol binge. On immune cells, acute alcohol intake seems to have dichotomous effects. On the one hand immunosuppressive and anti-inflammatory effects have been described, however, alcohol induced liver injury is driven by pro-inflammatory reactions. These immune effects seem to be driven by endotoxin or other bacterial products via Toll-like receptors that are translocated to the circulation via a defective gut barrier. Immune effects of alcohol have also been linked to hangover symptoms after an alcohol binge.

Furthermore there is evidence that endotoxemia might also contributes to alcohol dependence by promoting prolonged and increased voluntary alcohol intake in mice. On the other hand mutant mice lacking important genes for immune responses exhibit decreased alcohol consumption. This indicates that immune signaling promotes alcohol consumption. Therefore it is tempting to speculate that increased gut permeability leading to increased bacterial translocation after an acute alcohol binge could promote the desire for further alcohol consumption.

The investigators aim to test in this pilot trial whether one alcohol binge damages gut barrier function, increases bacterial translocation and causes innate immune dysfunction. Furthermore the effect of glucose and fructose will be studied too.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Age above 18 years
* Willingness to abstain from alcohol 48h prior to the study visits

Exclusion Criteria:

* Alcohol abuse .Alcohol Use Disorders Identification Test ≥ 8 in men or ≥ 7 in women or CAGE test ≥ 2 (both men and women)
* Elevated liver function test
* Any disease or medication that does not allow concomitant consumption of alcohol
* Women: pregnancy and lactation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers selected from a database
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Endotoxin assessed by percentage of endotoxin positive subjects | 4 hours
  Endotoxin measured by a HEK-blue cell based assay

SECONDARY OUTCOMES:
gut permeability (zonulin in stool) | 4 hours
  changes in gut permeability
bacterial translocation (bacterial DNA in serum) | 4 hours
  changes in bacterial translocation
oxidative stress (advanced oxidation protein products) | 4 hours
  changes in oxidative stress
inflammation (neutrophil oxidative burst) | 4 hours
  changes in inflammation
neutrophil phagocytic capacity | 4 hours
  changes in neutrophil function
gut microbiome composition | 4 hours
  changes in gut microbiome composition
fibroblast growth factor 21 (FGF21) | 4 hours
  changes in FGF21 serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria